CLINICAL TRIAL: NCT01499368
Title: A Multi-center, Randomized, Double-blind Phase III Clinical Trial to Assess and Compare to the Efficacy and Safety of Lafutidine, Famotidine and Omeprazole-referenced in Koran Erosive Esophagitis Patients
Brief Title: A Multi-center, Randomized, Double-blind Phase III Clinical Trial to Assess and Compare to the Efficacy and Safety of Lafutidine, Famotidine and Omeprazole-referenced in Korean Erosive Esophagitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAF-BR-CT-302
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — lafutidine; Famotidine; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lafutidine (Experimental): Lafutidine 20mg/day
  Interventions: Drug: Lafutidine
- Famotidine (Active Comparator): Famotidine 40mg/day
  Interventions: Drug: Famotidine
- Omeprazole (Other): Omeprazole 20mg/day
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Lafutidine — Lafutidine 20mg/day
  Arms: Lafutidine
Drug: Famotidine — Famotidine 40mg/day
  Arms: Famotidine
Drug: Omeprazole — Omeprazole 20mg/day
  Arms: Omeprazole

SUMMARY:
To evaluate the healing rate and safety of Lafutidine in erosive esophagitis

ELIGIBILITY:
Inclusion Criteria:

* Patients who had symptoms of heartburn with a diagnosis of grade A to D reflux esophagitis according to the Los Angeles classification

Exclusion Criteria:

* Gastric or duodenal ulcers (excluding ulcer scars)
* Concurrent presence of Barrett's esophagus
* A history of a poor response to H2RA or PPI given in the recommended dose for 8 weeks
* Other conditions considered by the attending physician to potentially affect the assessment of efficacy and safety

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Woo Lee, Study Chair — Korea University Ansan Hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- Lafutidine: Lafutidine 20mg/day
  Lafutidine 10mg bid, po
- Famotidine: Famotidine 40mg/day
  Famotidine 20mg bid, po
- Omeprazole: Omeprazole 20mg/day
  Omeprazole 20mg qd(daily), po
Period: Overall Study
Arm/Group | Lafutidine | Famotidine | Omeprazole
Started | 165 | 163 | 167
Completed | 138 | 145 | 146
Not Completed | 27 | 18 | 21
Not completed — Did not meet I/E criteria | 8 | 4 | 4
Not completed — Prohibited Concomitant medication | 1 | 1 | 0
Not completed — Withdrawal by Subject | 11 | 10 | 8
Not completed — Lost to Follow-up | 3 | 2 | 5
Not completed — Adverse Event | 4 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Deviation from visit window | 0 | 0 | 1
Not completed — Error of Prescriptions | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Because of a Duplicated subject in Active comparator, One was excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lafutidine | Famotidine | Omeprazole | Total
Number analyzed (Participants) | 165 | 162 | 167 | 494
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age, Mean+-STD (years) | 50.20 (13.57) | 51.25 (12.76) | 49.65 (13.84) | 50.36 (13.39)
Age, Continuous [Median (Full Range); unit: years] | 53.00 [21.00 to 73.00] | 53.00 [24.00 to 74.00] | 50.00 [20.00 to 74.00] | 52.00 [20.00 to 74.00]
Age, Customized [Count of Participants; unit: Participants]
  20 years~ 29 years | 18 | 10 | 16 | 44
  30 years ~ 39 years | 22 | 23 | 30 | 75
  40 years ~ 49 years | 25 | 30 | 32 | 87
  50 years ~ 59 years | 55 | 49 | 41 | 145
  60 years ~ 69 years | 36 | 40 | 37 | 113
  70 years ~ 74 years | 9 | 10 | 11 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 48 | 46 | 154
  Male | 105 | 114 | 121 | 340

OUTCOME MEASURES:

1. Primary Outcome: Recovery Rates of Reflux Esophagitis
Description: Recovery rates of reflux esophagitis on the Esophago Gastro Duodenoscopy test after 8 week treatment-FAS
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lafutidine | Famotidine | Omeprazole
Number analyzed (Participants) | 144 | 145 | 147
Participants
  Recovered | 101 | 92 | 126
  Not recovered | 43 | 53 | 21
Statistical Analysis 1: Comparison: Lafutidine vs Famotidine; Test type: Non-Inferiority — Non-inferiority: The Lower limit is not lower than -15%; p = 0.05, Chi-squared

2. Secondary Outcome: The Proportion of Days Without 'Cardinal Symptom'
Description: The proportion of days without 'Cardinal symptom' after 4 or 8 week treatment-FAS 'Cardinal symptom': Burning sesation in the chest, Acid reflux, Heartburn including chest pain
Time Frame: 4 or 8 week
Population: Missing = Lafutidine(5) , Omeprazole(1)
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Lafutidine | Famotidine | Omeprazole
Number analyzed (Participants) | 139 | 145 | 146
proportion of days
  week 4 | 0.64 (0.31) | 0.56 (0.32) | 0.69 (0.30)
  week 8: number analyzed (Participants) | 139 | 144 | 146
  week 8 | 0.77 (0.27) | 0.67 (0.32) | 0.82 (0.24)
  week 8(LOCF) | 0.77 (0.27) | 0.67 (0.32) | 0.82 (0.24)
Statistical Analysis 1: Comparison: Lafutidine vs Famotidine; Test type: Non-Inferiority — Non-Inferiority; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test

3. Secondary Outcome: The Proportion of Daytimes Without 'Cardinal Symptom'
Description: The proportion of daytimes without 'Cardinal symptom' after 4 or 8 week treatment-FAS 'Cardinal symptom': Burning sensation in the chest, Acid reflux, Heartburn including chest pain
Time Frame: 4 or 8 week
Population: Missing = Lafutidine(5) , Omeprazole(1)
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Lafutidine | Famotidine | Omeprazole
Number analyzed (Participants) | 139 | 145 | 146
proportion of days
  week 4 | 0.74 (0.27) | 0.68 (0.29) | 0.77 (0.27)
  week 8: number analyzed (Participants) | 139 | 144 | 146
  week 8 | 0.83 (0.23) | 0.76 (0.28) | 0.87 (0.20)
  week 8(LOCF) | 0.83 (0.23) | 0.76 (0.28) | 0.87 (0.20)

4. Secondary Outcome: The Proportion of Nighttimes Without 'Cardinal Symptom'
Description: The proportion of Nighttimes without 'Cardinal symptom' after 4 or 8 treatment-FAS 'Cardinal symptom': Burning sensation in the chest, Acid reflux, Heartburn including chest pain
Time Frame: 4 or 8 week
Population: Missing = Lafutidine(5) , Omeprazole(1)
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Lafutidine | Famotidine | Omeprazole
Number analyzed (Participants) | 139 | 145 | 146
proportion of days
  week 4 | 0.75 (0.27) | 0.72 (0.30) | 0.82 (0.23)
  week 8: number analyzed (Participants) | 139 | 144 | 146
  week 8 | 0.87 (0.19) | 0.78 (0.29) | 0.89 (0.18)
  week 8(LOCF) | 0.87 (0.19) | 0.78 (0.29) | 0.89 (0.18)

ADVERSE EVENTS:
Time Frame: 4 week, 8 week and 9 week
Arm/Group | Lafutidine | Famotidine | Omeprazole
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/162 | 3/167
Other Adverse Events (participants affected / at risk) | 36/165 | 30/162 | 34/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lafutidine (N=165) | Famotidine (N=162) | Omeprazole (N=167)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — During the treatment period, he got biopsy at the Dermatology for skin lesion on the left inguinal area, which he had 2 years ago. The result was basal cell carcinoma, but the physician judged that causality of this event with the IP was unlikely.
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — He had musculoskeletal pain because of a car accident, during the treatment period. The physician confirmed that this shoulder pain was caused by muscle tears, which he originally had, and judged that causality of this event with IP was unlikely.
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) — Pregnancy After 1 month of the treatment peroid, she dropped out of the trial. About 7 months later, she gave birth to a healthy baby boy.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lafutidine (N=165) | Famotidine (N=162) | Omeprazole (N=167)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (10) | 2 (3) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Acute pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Mixed incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No